CLINICAL TRIAL: NCT05249049
Title: An Osseointegrated Transtibial Prosthesis Offering Long-Term Bi-Directional Efferent-Afferent Neural Transmission
Brief Title: Osseointegrated Transtibial Prosthesis With Neural Interface
Acronym: TTeOPRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts Institute of Technology (Other)
Collaborators: Brigham and Women's Hospital (Other); Integrum (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012000283
Record Dates: First submitted 2021-12-03; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Amputation
Keywords: Osseointegration; Prosthesis; Neural Transmission

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- e-OPRA Implant System for Transtibial Amputees (Experimental): Implantation of e-OPRA Implant System in lower limb.
  Interventions: Device: e-OPRA Implant System for Transtibial Amputees

INTERVENTIONS:
Device: e-OPRA Implant System for Transtibial Amputees — The e-OPRA System for transtibial use consists of an anchorage element (Fixture), which is surgically inserted in the medullary canal of the amputated skeleton of the lower limb. The skin penetrating e-Abutment is then inserted and secured with the e-Abutment screw. To allow the system to be used with an external neuro-mechanical prosthesis, soft tissues from the distal limb are preserved incorporated into the residual limb. Muscle electrodes are then placed in the neuro-muscular constructs. After a rehabilitation program, in everyday use, the implanted e-OPRA device will be used by the patient with the Axor TC and their commercially available prosthesis. However, the modified version of the implant will allow the patient to use a powered neuro-mechanical prosthesis during specified testing scenarios.
  Other Names: e-OPRA

SUMMARY:
The e-OPRA Implant System, is a further development of the OPRA (Osseointegrated Prostheses for the Rehabilitation of Amputees) Implant System. The e-OPRA Implant system is an implant system for direct skeletal anchorage of amputation prostheses. The added feature in the e-OPRA Implant system, is a bidirectional interface into the human body that allows permanent and reliable communication using implanted electrodes. These electrodes will provide long-term stable bioelectric signals for an improved control of the prosthetic limb. The purpose of the study is to evaluate the feasibility of a transtibial amputee with the e-OPRA Implant System exhibiting full neural control over a neuro-mechanical prosthetic system.

A maximum of two subjects will be enrolled. Each subject will undergo a surgery where the e-OPRA Implant System will be implanted. The subjects will participate in follow-up sessions of which the last one occurs approximately 24 months after the surgery. This is a prospective, non-randomized, uncontrolled study.

DETAILED DESCRIPTION:
Normalization of function for individuals with limb amputation is within reach, and will be achieved by smart implants capable of bi-directional communication between brain and machine via bone-anchored, interactive, powered prosthetic components. Rehabilitation of patients with expected high physical activity level, such as after amputation due to trauma or cancer, is currently limited by dependence on an external socket for the mechanical attachment of the prosthesis to the residuum. Despite the use of advanced materials and fabrication methods, socket interfaces routinely cause sores, chafing, pain, increased energy expenditure, and a decreased quality of life. Novel surgical techniques using osseointegrated transdermal titanium implants, now validated in Europe for 25 years, obviate the need for painful sockets by establishing a direct, load-bearing link between skeleton and prosthesis. This system also promises a transformative breakthrough in neuroprosthetics, because it allows for fully internal, high bandwidth, stable neural connections. In a paper recently published in Science Translational Medicine, implanted muscle and nerve cuff electrodes were added to the osseointegrated device, creating a bi-directional efferent-afferent interface utilizing a safe and immune-sealed osseo-conduit. Commenting on this work, the editor stated, "Osseointegration could revolutionize the field of neuroprosthetics, giving patients more intuitive control and more freedom of movement."

Investigators have sought to advance bionic prostheses with sufficient degrees of freedom for performing natural tasks, such as manipulating objects in the case of upper-extremity prostheses, or walking and running for lower-extremity systems. Nonetheless, afferent feedback has not played a major role in any clinically-viable amputation prostheses, despite being critical for biomimetic control. This deficiency can, in large part, be attributed to a lack of clinically-available methodologies for sustained communication with the peripheral nervous system. There is no existing platform capable of invasive, robust, and permanent communication with the peripheral nervous system in a high-demand clinical setting. Only by bringing together critical technologies and expertise will it be possible to create a bionic limb replacement system with adequate suspension, load transmission, motor control, proprioceptive feedback, and external mechatronics that resemble the mass, volume and dynamics of the missing biological limb.

To achieve such an unprecedented integration of prosthetic technology, a broad scientific team has been assembled with members from Massachusetts Institute of Technology (MIT: Carty, Herr, Riso, Braanemark), Brigham and Women's Hospital (BWH: Carty), University of California, San Francisco (UCSF: O'Donnell), University of Michigan (U-M: Cederna), and Walter Reed National Military Medical Center (WRNMMC: Forsberg, Potter). With this combination of leading technologists and clinicians in the fields of biomechanics, osseointegration, prosthetics, implantable electrodes, sensory feedback, proprioception, reconstructive surgery, and mechatronics, we seek to develop the most advanced clinically-viable artificial limb. With proprioceptive afferent feedback, we seek to demonstrate that a person with transtibial amputation can exhibit full volitional control over a neuro-mechanical prosthetic system where key walking metrics are normalized, including preferred speed, metabolism and joint dynamics. It is the view of the proposers that the scope of this research is fundamental wherein the results will be shared broadly within the scientific community.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female age 22-65 at the time of surgery.
* The patient must have an existing unilateral or bilateral transtibial amputation or a medical condition requiring performance of a unilateral or bilateral transtibial amputation with a minimum of 8 cm of residual tibia after amputation.
* The subject must have undergone independent consultation with at least two lower extremity surgical specialists to ensure they have exhausted all limb salvage options prior to undergoing amputation, as well as a psychiatric evaluation to ensure appropriate capacity and volition.
* The patient must have the ability to ambulate at variable cadence (an expected lower extremity prosthesis functional level of K3 or above).
* The patient must have adequate bone stock to support the implanted device.
* The patient must have adequate soft tissue bulk and muscle mass present in the operative limb to support appropriate wound healing and muscle end organ construction.
* In the opinion of the investigator, normal cognitive function and absence of any physical limitations, addictive diseases or underlying medical conditions that may preclude patient from being a good surgical and/or study candidate.
* Willingness, ability and commitment to participate in baseline and follow-up evaluations for the full length of the study including the prescribed rehabilitation program.
* Written informed consent to participate in the study provided by the patient or legal representative.

Exclusion Criteria:

* Women who are pregnant, lactating or planning a pregnancy during the first twelve (12) months of the post-surgical follow-up.
* Subjects who have not been completely abstinent from tobacco use for at least 6 weeks preoperatively.
* Subjects who weigh over 90 kg.
* Subjects who have an active infection or dormant bacteria.
* Subjects would have less than 2 mm of remaining cortex bone available around the implant, if implanted.
* Subjects with advanced atrophic muscle and and/or compromised soft tissue coverage in the operative limb.
* Evidence of or a documented history of severe peripheral vascular disease, diabetes mellitus (type I or type II), skin diseases, Neuropathy or neuropathic disease and severe phantom pain, or osteoporosis, such that, in the opinion of the investigator, will not allow the subject to be a good study candidate.
* Evidence of any active skin disease involving the proposed surgical limb.
* History of systemically administered corticosteroids, immune-suppressive therapy or chemotherapy drugs within six (6) months of implant surgery.
* Severe co-morbidity, atypical skeletal anatomy, or poor general physical/mental health that, in the opinion of the Investigator, will not allow the subject to be a good study candidate (i.e. other disease processes, mental capacity, substance abuse, shortened life expectancy, vulnerable patient population, BMI >40, etc.).
* The subject is currently involved in another clinical study where that participation may conflict or interfere with the treatment, follow-up or results of this clinical study.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-04-15 (Estimated)

PRIMARY OUTCOMES:
Electrode Robustness and Connector/Lead Integrity (resistance) | 24 months
  Measured Impedance of electrode(kOhms)
Electrode Robustness and Connector/Lead Integrity (amplitude) | 24 months
  Maximal Voluntary Contraction Amplitude (mV)
Sensor Function and Signal Quality | 24 months
  Signal-to-noise ratio (SNR) above 2

SECONDARY OUTCOMES:
Preferred Walking Speed | 24 months
  Preferred walking speed, as each subject ambulates with the neuromechanical prosthesis, will be evaluated. Preferred walking speed will be compared to a non-amputee height/weight match for each enrolled subject. A baseline data set will first be collected for each subject ambulating with a conventional prosthesis. Each subject will be timed as they traverse a predetermined distance at a steady speed that they deem most comfortable.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - MIT Media Lab, Cambridge, Massachusetts